CLINICAL TRIAL: NCT01191944
Title: A Double-blind, Double-dummy, Randomised, Parallel-group Study Comparing the Efficacy, Safety and Tolerability of Pramipexole Extended Release Versus Pramipexole Immediate Release Administered Orally for 18 Weeks in Chinese Parkinson's Disease (PD) Patients Who Can be Concomitantly Treated With Levodopa
Brief Title: Pramipexole Extended Release Versus Pramipexole Immediate Release for 18 Weeks in Chinese Parkinson's Disease (PD) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 248.671
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- pramipexole Extended release (Experimental): subjects will receive 0.375mg once a day to 4.5mg once a day depending on investigator's judgement
  Interventions: Drug: pramipexole extended release tablet
- pramipexole Immediate release (Active Comparator): subjects will receive 0.125mg three times a day to 1.0mg three times a day depending on investigator's judgement
  Interventions: Drug: pramipexole immediate release tablet

INTERVENTIONS:
Drug: pramipexole immediate release tablet — 0.375mg-4.5mg(daily dose), three times a day
  Arms: pramipexole Immediate release
Drug: pramipexole extended release tablet — 0.375mg-4.5mg, once a day
  Arms: pramipexole Extended release

SUMMARY:
The objective of this trial is to evaluate non-inferiority of pramipexole Extended release to Immediate release at 18 weeks on the primary efficacy endpoint (Unified Parkinson's Disease Rating Scale II+III) in Chinese PD patients who can be concomitantly treated with Levodopa .

ELIGIBILITY:
Inclusion criteria:

1. Male or female Chinese patient with idiopathic Parkinson's disease (PD) confirmed by at least two of the following signs: resting tremor, bradykinesia, rigidity.
2. Parkinson's disease diagnosed for at least 2 years.
3. Patients 30 years of age or older at the time of diagnosis.
4. Modified Hoehn and Yahr stage of 2 to 4 at on-time.
5. If a patient is treated with standard or controlled release Levodopa combined with a Dopa-Decarboxylase-inhibitor or with Levodopa combined with a Dopa-Decarboxylase-inhibitor/entacapone, the dosage should be optimised according to investigator's judgement, and stable for at least 4 weeks prior to baseline visit.
6. If a patient treated with Levodopa combined with a Dopa-Decarboxylase-inhibitor has motor fluctuations, he should not have more than 6 hours of off-time every day during waking hours (documented on a patient diary completed for 2 consecutive days before baseline visit).
7. Patient willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures (in particular, after training, the patient should be able to recognise the off-time and on-time periods during waking hours and to record them accurately in the patient diary).
8. Signed informed consent obtained before any study procedures are carried out (in accordance with International Conference on Harmonisation-Good Clinical Practice guidelines and local legislation).

Exclusion criteria:

Medical exclusions:

1. Atypical parkinsonian syndromes due to drugs (e.g., metoclopramide, flunarizine), metabolic disorders (e.g., Wilson's disease), encephalitis or degenerative diseases (e.g., progressive supranuclear palsy).
2. Dementia, as defined by a Mini-Mental State Exam score < 24 at screening visit [R96-2656].
3. Any psychiatric disorder according to Diagnostic and Statistical Manual of Mental Disorders (4th edition)criteria that could prevent compliance or completion of the study and/or put the patient at risk if he/she takes part in the study.
4. History of psychosis, except history of drug induced hallucinations (provided the investigator considers that participation to the trial would not represent a significant risk for the patient).
5. History of deep brain stimulation
6. Clinically significant electrocardiogram abnormalities at screening visit, according to investigator's judgement.
7. Clinically significant hypotension (i.e. supine systolic blood pressure < 90 mmHg) and/or symptomatic orthostatic hypotension (i.e. clinical symptoms of orthostatic hypotension associated with a decline >=20 mmHg in systolic blood pressure and a decline >= 10 mmHg in diastolic blood pressure, at one minute after standing compared with the previous supine systolic and diastolic blood pressure obtained after 5 minutes of quiet rest) at screening or baseline visit.
8. Malignant melanoma or history of previously treated malignant melanoma.
9. Any other clinically significant disease, whether treated or not, that could put the patient at risk or could prevent compliance or completion of the study.
10. Pregnancy (to be excluded by urine pregnancy test at screening visit) or breast-feeding.
11. Sexually active female of childbearing potential (less than 6 months post-menopausal and not surgically sterilised) not using a medically approved method of birth control (i.e. oral contraceptives, intrauterine device, or double-barrier) for at least one month prior to the screening visit and throughout the study period (up to the follow-up visit).
12. Serum levels of Aspartate Aminotransferase, Alanine Aminotransferase , alkaline phosphatases or total bilirubin > 2 Upper Limit of Normal (on screening lab test).
13. Patients with a creatinine clearance < 50 mL/min/1.73m2 (estimated by the local lab / the investigator using the Modification of Diet in Renal Disease (MDRD), and calculated on screening lab test)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (20):
- China (20):
  - 248.671.86004 Boehringer Ingelheim Investigational Site, Beijing
  - 248.671.86006 Boehringer Ingelheim Investigational Site, Beijing
  - 248.671.86007 Boehringer Ingelheim Investigational Site, Beijing
  - 248.671.86020 Boehringer Ingelheim Investigational Site, Beijing
  - 248.671.86012 Boehringer Ingelheim Investigational Site, Chengdu
  - 248.671.86013 Boehringer Ingelheim Investigational Site, Chongqing
  - 248.671.86014 Boehringer Ingelheim Investigational Site, Chongqing
  - 248.671.86008 Boehringer Ingelheim Investigational Site, Guangzhou
  - 248.671.86009 Boehringer Ingelheim Investigational Site, Guangzhou
  - 248.671.86017 Boehringer Ingelheim Investigational Site, Hangzhou
  - 248.671.86018 Boehringer Ingelheim Investigational Site, Hangzhou
  - 248.671.86005 Boehringer Ingelheim Investigational Site, Jinan
  - 248.671.86002 Boehringer Ingelheim Investigational Site, Nanjing
  - 248.671.86001 Boehringer Ingelheim Investigational Site, Shanghai
  - 248.671.86003 Boehringer Ingelheim Investigational Site, Shanghai
  - 248.671.86010 Boehringer Ingelheim Investigational Site, Shanghai
  - 248.671.86011 Boehringer Ingelheim Investigational Site, Shenyang
  - 248.671.86019 Boehringer Ingelheim Investigational Site, Suzhou
  - 248.671.86015 Boehringer Ingelheim Investigational Site, Wuhan
  - 248.671.86016 Boehringer Ingelheim Investigational Site, Wuhan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Whilst 475 patients were enrolled only 473 were treated, since one patient was not compliant to protocol and did not take any trial drug and another refused to take trial medication.
Groups:
- Pramipexole ER: Pramipexole Extended Release (ER). Tablets of 0.375 mg and 1.5 mg administered once daily (qd) to achieve daily doses of 0.375 mg, 0.75 mg, 1.5 mg, 2.25 mg, 3.0 mg, 3.75 mg or 4.5 mg
- Pramipexole IR: Pramipexole Immediate Release (IR). Tablets of 0.125 mg, 0.25 mg and 1.0 mg administered 3 times daily to achieve a total daily dose of 0.375 mg, 0.75 mg, 1.5 mg, 2.25 mg, 3.0 mg, 3.75 mg, or 4.5 mg
Period: Overall Study
Arm/Group | Pramipexole ER | Pramipexole IR
Started | 234 (Treated titration/maintenance) | 239 (Treated titration/maintenance)
Completed | 217 (Completed titration/maintenance) | 220 (Completed titration/maintenance)
Not Completed | 17 | 19
Not completed — Adverse Event | 11 | 12
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Population: Treated Set, all randomized patients that received treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Pramipexole ER | Pramipexole IR | Total
Number analyzed (Participants) | 234 | 239 | 473
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.10) | 61.8 (9.03) | 62.0 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 95 | 175
  Male | 154 | 144 | 298

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Unified Parkinsons Disease Rating Scale (UPDRS) Parts II+III Score at Week 18
Description: UPDRS total score ranges from 0 (best) to 160 (worst) and was calculated as the sum of Part II (activities of daily living, ranges from 0 to 52) and Part III (motor examination, ranges from 0 to 108). Reduction over time represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: Full analysis set (FAS) with last observation carried forward (LOCF). FAS is defined as all randomised patients which received at least one dose of study drug and provided any post baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 228 | 236
Units on a scale | -13.807 (0.6547) | -13.047 (0.6434)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; The null hypothesis (H0) states that the mean change from baseline to Week 18 (or last observation carried forward [LOCF]) in the UPDRS II+III score for the treatment group pramipexole ER is inferior to the mean change for the treatment group pramipexole IR; Test type: Non-Inferiority or Equivalence — pre-specified non-inferiority (NI) margin of -4 points; p < 0.0001, ANCOVA — one-sided test relative to NI margin of -4; adjusted for treatment, centre and baseline; Mean Difference (Final Values) = 0.760, 95% CI [-1.047 to 2.566], Standard Error of Mean 0.9192 — Pramipexole IR minus Pramipexole ER, Pramipexole ER non inferior to Pramipexole IR if lower limit of confidence interval (CI) for the mean difference is higher than NI margin

2. Secondary Outcome: Change From Baseline in Percentage Off-time During Waking Hours at Week 18
Description: Percentage off-time during waking hours based on patient diary data, percentage ranging from 0 (best case) to 100 (worst case). Off-time describes a period when the patient experiences increased parkinsonian symptoms (e.g. immobility or inability to move with ease). Reduction over time represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: FAS (LOCF) reduced to patients with advanced Parkinsons Disease (PD). Advanced PD patients were those reporting at least 2 hours of off-time daily during each of the two days before baseline, as recorded in the patient diary.
Measure: Least Squares Mean (Standard Error); unit: Percentage off-time
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 110 | 106
Percentage off-time | -6.962 (1.5072) | -7.443 (1.5362)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.8261, ANCOVA; Mean Difference (Final Values) = -0.480, 95% CI 2-sided [-4.787 to 3.826], Standard Error of Mean 2.1836

3. Secondary Outcome: Change From Baseline in Duration of Off-time During Waking Hours at Week 18
Description: Duration of off-time during waking hours based on patient diary data. Off-time describes a period when the patient experiences increased parkinsonian symptoms (e.g. immobility or inability to move with ease). Reduction over time represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: FAS (LOCF) reduced to patients with advanced PD. Advanced PD patients were those reporting at least 2 hours of off-time daily during each of the two days before baseline, as recorded in the patient diary.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 110 | 106
hours | -1.044 (0.2256) | -1.098 (0.2300)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.8698, ANCOVA; Mean Difference (Final Values) = -0.054, 95% CI 2-sided [-0.699 to 0.592], Standard Error of Mean 0.3274

4. Secondary Outcome: Responder in Percentage Off-time During Waking Hours at Week 18
Description: Percentage off-time based on patient diary data, percentage ranging from 0 (best case) to 100 (worst case). Off-time describes a period when the patient experiences increased parkinsonian symptoms (e.g. immobility or inability to move with ease). Reduction over time represents an improvement. Responders were defined as patients with at least a 20 percent improvement relative to baseline.
Time Frame: Baseline and week 18
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 110 | 106
Participants
  Responder | 58 | 59
  Non-Responder | 52 | 47
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.7902, Cochran-Mantel-Haenszel

5. Secondary Outcome: Change From Baseline in Percentage On-time Without Dyskinesia at Week 18
Description: Percentage on-time without Dyskinesia based on patient diary data, percentage ranging from 0 (worst case) to 100 (best case). On-time describes a period during which a patient was relatively free of Parkinsons symptoms (e.g. mobile or capable of moving with relative ease and independence). Increase in the percentage represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of on-time
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 110 | 106
Percentage of on-time | 7.028 (1.9274) | 4.265 (1.9643)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.3223, ANCOVA; Median Difference (Final Values) = -2.763, 95% CI 2-sided [-8.255 to 2.729], Standard Error of Mean 2.7845

6. Secondary Outcome: Change From Baseline in Percentage On-time With Non-troublesome Dyskinesia at Week 18
Description: Percentage on-time with non-troublesome Dyskinesia based on patient diary data, percentage ranging from 0 (worst case) to 100 (best case). On-time describes a period during which a patient was relatively free of Parkinsons symptoms (e.g. mobile or capable of moving with relative ease and independence). Dyskinesia qualified as non-troublesome if it did not interfere with function or did not cause meaningful discomfort. Increase in the percentage represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of on-time
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 110 | 106
Percentage of on-time | -0.235 (1.0807) | 3.275 (1.1013)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.0254, ANCOVA; Mean Difference (Final Values) = 3.510, 95% CI 2-sided [0.437 to 6.583], Standard Error of Mean 1.5581

7. Secondary Outcome: Change From Baseline in Percentage On-time Without or With Non-troublesome Dyskinesia at Week 18
Description: Percentage on-time without or with non-troublesome Dyskinesia based on patient diary data, percentage ranging from 0 (best case) to 100 (worst case). On-time describes a period during which a patient was relatively free of Parkinsons symptoms (e.g. mobile or capable of moving with relative ease and independence). Dyskinesia qualified as non-troublesome if it did not interfere with function or did not cause meaningful discomfort. Increase in the percentage represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of on-time
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 110 | 106
Percentage of on-time | 6.855 (1.5672) | 7.476 (1.5973)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.7843, ANCOVA; Mean Difference (Final Values) = 0.621, 95% CI 2-sided [-3.848 to 5.090], Standard Error of Mean 2.2658

8. Secondary Outcome: Change From Baseline in Percentage On-time With Troublesome Dyskinesia at Week 18
Description: Percentage on-time with troublesome Dyskinesia based on patient diary data, percentage ranging from 0 (best case) to 100 (worst case). On-time describes a period during which a patient was relatively free of Parkinsons symptoms (e.g. mobile or capable of moving with relative ease and independence). Dyskinesia qualified as troublesome if it interfered with function or caused meaningful discomfort. Decrease in the percentage represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of on-time
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 110 | 106
Percentage of on-time | -0.142 (0.3398) | 0.226 (0.3463)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.4529, ANCOVA; Median Difference (Final Values) = 0.369, 95% CI 2-sided [-0.598 to 1.335], Standard Error of Mean 0.4901

9. Secondary Outcome: Change From Baseline in Duration of On-time Without Dyskinesia at Week 18
Description: Duration of on-time without Dyskinesia based on patient diary data. On-time describes a period during which a patient was relatively free of Parkinsons symptoms (e.g. mobile or capable of moving with relative ease and independence). Increase in the duration represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 110 | 106
hours | 1.026 (0.3076) | 0.496 (0.3134)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.2338, ANCOVA; Mean Difference (Final Values) = -0.530, 95% CI 2-sided [-1.405 to 0.345], Standard Error of Mean 0.4437

10. Secondary Outcome: Change From Baseline in Duration of On-time With Non-troublesome Dyskinesia at Week 18
Description: Duration on-time with non-troublesome Dyskinesia based on patient diary data, percentage ranging from 0 (worst case) to 100 (best case). On-time describes a period during which a patient was relatively free of Parkinsons symptoms (e.g. mobile or capable of moving with relative ease and independence). Dyskinesia qualified as non-troublesome if it did not interfere with function or did not cause meaningful discomfort. Increase in the duration represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 110 | 106
hours | -0.044 (0.1740) | 0.518 (0.1773)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.0263, ANCOVA; Mean Difference (Final Values) = 0.562, 95% CI 2-sided [0.067 to 1.057], Standard Error of Mean 0.2509

11. Secondary Outcome: Change From Baseline in Duration of On-time Without or With Non-troublesome Dyskinesia at Week 18
Description: Duration of on-time without Dyskinesia or with non-troublesome Dyskinesia based on patient diary data, percentage ranging from 0 (worst case) to 100 (best case). On-time describes a period during which a patient was relatively free of Parkinsons symptoms (e.g. mobile or capable of moving with relative ease and independence). Dyskinesia qualified as non-troublesome if it did not interfere with function or did not cause meaningful discomfort. Increase in the duration represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 110 | 106
hours | 0.982 (0.2583) | 1.013 (0.2632)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.9337, ANCOVA; Mean Difference (Final Values) = 0.031, 95% CI 2-sided [-0.704 to 0.766], Standard Error of Mean 0.3727

12. Secondary Outcome: Change From Baseline in Duration of On-time With Troublesome Dyskinesia at Week 18
Description: Duration of on-time with troublesome Dyskinesia based on patient diary data, percentage ranging from 0 (best case) to 100 (worst case). On-time describes a period during which a patient was relatively free of Parkinsons symptoms (e.g. mobile or capable of moving with relative ease and independence). Dyskinesia qualified as troublesome if it interfered with function or caused meaningful discomfort. Decrease in the duration represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 110 | 106
hours | -0.000 (0.0553) | 0.031 (0.0564)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.6995, ANCOVA; Mean Difference (Final Values) = 0.031, 95% CI 2-sided [-0.127 to 0.188], Standard Error of Mean 0.0798

13. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Responder at Week 18
Description: CGI-I was used to assess the overall status of Parkinsons disease (PD) after interviewing the patient about the various aspects of the PD and after evaluating adverse events and concomitant treatments. Ranging from 1 point=very much improved to 7 points=very much worse. Responders were defined as patients having score 1 or 2 (at least much improved) when comparing the past week to the assessment at baseline.
Time Frame: 18 weeks
Population: FAS (LOCF). Only patients with on-treatment CGI-I evaluation were analyzed.
Measure: Number; unit: Participants
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 224 | 233
Participants
  Responder | 125 | 138
  Non-Responder | 99 | 95
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.3170, Cochran-Mantel-Haenszel

14. Secondary Outcome: Patient Global Impressions of Improvement (PGI-I) Responder at Week 18
Description: The PGI-I scale is a patient-rated instrument which was used to measure the improvement of a patients PD symptoms throughout the study. Ranging from 1 point=very much better to 7 points=very much worse. Responders were defined as patients having score 1 or 2 (at least much better) when comparing the past week to the assessment at baseline.
Time Frame: 18 weeks
Population: FAS (LOCF)
Measure: Number; unit: Participants
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 228 | 236
Participants
  Responder | 119 | 127
  Non-Responder | 109 | 109
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.4756, Cochran-Mantel-Haenszel

15. Secondary Outcome: Responder in UPDRS Parts II+III Score at Week 18
Description: Responders were defined as patients with at least a 20 percent improvement of UPDRS II+III score relative to baseline. UPDRS II+III ranges 0-160 scores from best to worst and was calculated as the sum of Part II (activities of daily living, ranges from 0 to 52) and Part III (motor examination, ranges from 0 to 108).
Time Frame: Baseline and week 18
Population: FAS (LOCF)
Measure: Number; unit: Participants
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 228 | 236
Participants
  Responder | 164 | 154
  Non-Responder | 64 | 82
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.1051, Cochran-Mantel-Haenszel

16. Secondary Outcome: Change From Baseline in UPDRS II Score Separately at Week 18
Description: UPDRS Part II (activities of daily living) ranges from 0 to 52. Reduction over time represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: FAS (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 228 | 236
Units on a scale | -3.750 (0.2235) | -3.596 (0.2197)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.6237, ANCOVA; Mean Difference (Final Values) = 0.154, 95% CI 2-sided [-0.463 to 0.771], Standard Error of Mean 0.3138

17. Other Pre Specified Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Total Score at 18 Weeks
Description: ESS is a patient-report scale with 8 items rating how likely one is to fall asleep during passive and inconsequential situations such as watching television, more active situations such as sitting and talking to someone, or consequential situations such as sitting in a car, while stopped for a few minutes in traffic. The likelihood of dozing off is rated from 0 points (no chance) to 3 points (high chance). The overall rating scale is scored from 0 (no daytime sleep) to 24 (worst daytime sleep).
Time Frame: Baseline and week 18
Population: Observed cases (OC). Only patients with ESS assessment at baseline and at 18 weeks were analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 217 | 215
Units on a scale | 0.1 (3.43) | -0.0 (3.38)

18. Secondary Outcome: Change From Baseline in UPDRS III Score Separately at Week 18
Description: UPDRS Part III (motor examination) ranges from 0 to 108. Reduction over time represents an improvement. Means are adjusted for treatment, centre and baseline.
Time Frame: Baseline and week 18
Population: FAS (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 228 | 236
Units on a scale | -10.068 (0.5048) | -9.440 (0.4962)
Statistical Analysis 1: Comparison: Pramipexole ER vs Pramipexole IR; Test type: Superiority or Other; p = 0.3760, ANCOVA; Mean Difference (Final Values) = 0.628, 95% CI 2-sided [-0.765 to 2.021], Standard Error of Mean 0.7088

19. Secondary Outcome: Levodopa (L-Dopa) Introduction During the Study
Description: Number of patients without concomitant L-Dopa treatment at baseline which required L-Dopa supplementation during the study.
Time Frame: 18 weeks
Population: FAS. Only patients without concomitant L-Dopa treatment at baseline.
Measure: Number; unit: Participants
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 25 | 40
Participants
  with L-Dopa introduction | 1 | 0
  without L-Dopa introduction | 24 | 40

20. Secondary Outcome: Levodopa (L-Dopa) Dose Change During the Study
Description: Although the number of patients who began the study with concomitant L-dopa supplementation and required a change in dosage was not analysed for this study, the change from baseline in L-dopa dose is presented.
Time Frame: 18 weeks
Population: FAS. Only patients with concomitant L-Dopa treatment at baseline.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Pramipexole ER | Pramipexole IR
Number analyzed (Participants) | 203 | 196
mg | -5.17 (51.563) | -11.22 (101.913)

ADVERSE EVENTS:
Time Frame: Up to 18 weeks
Arm/Group | Pramipexole ER | Pramipexole IR
Serious Adverse Events (participants affected / at risk) | 6/234 | 13/239
Other Adverse Events (participants affected / at risk) | 93/234 | 90/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole ER (N=234) | Pramipexole IR (N=239)
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole ER (N=234) | Pramipexole IR (N=239)
Constipation (Gastrointestinal disorders) | 17 | 20
Nausea (Gastrointestinal disorders) | 20 | 17
Dizziness (Nervous system disorders) | 30 | 31
Dyskinesia (Nervous system disorders) | 12 | 18
Somnolence (Nervous system disorders) | 51 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.